CLINICAL TRIAL: NCT04496063
Title: USTekinumab in Fistulising Perianal Crohn's Disease (CD): The USTAP CD Study
Brief Title: USTekinumab in Fistulising Perianal Crohn's Disease (USTAP)
Acronym: USTAP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-2019-01
Record Dates: First submitted 2020-06-29; First posted 2020-08-03 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Fistulising Perianal; Placebo; Ustekinumab; Double-blind
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Ustekinumab (Experimental): Intravenous induction (6mg/kg) followed by Ustekinumab subcutaneous 90mg every 8 weeks
  Interventions: Drug: Ustekinumab
- Group 2 Placebo (Placebo Comparator): Placebo intravenous followed by Placebo subcutaneous every 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab — Intravenous induction (6mg/kg) followed by Ustekinumab subcutaneous 90mg every 8 weeks
  Other Names: Stelara
  Arms: Group 1 Ustekinumab
Drug: Placebo — Placebo intravenous followed by Placebo subcutaneous every 8 weeks
  Arms: Group 2 Placebo

SUMMARY:
Phase IV

Trial design : Multicentre, randomized, double-blind, placebo-controlled study

Population : Moderate to severe Crohn's disease with at least one active perianal fistula track

Investigational treatment : Group 1: Ustekinumab (UST) IntraVenous (IV) induction (6mg/kg) followed by UST SubCutaneous (SC) 90mg every 8 weeks. Group 2: Placebo IV followed by Placebo SC The trial duration for each patient will be 48 weeks.

Trial objective : To evaluate the efficacy and safety of ustekinumab in fistulizing perianal Crohn's disease.

Number of patients : A total of 146 patients will be included in 20 sites in France

Trial duration : First patient in: Q3 2020 - Last patient first visit: Q3 2022 Last patient last visit: Q3 2023

DETAILED DESCRIPTION:
Main endpoint:

The primary endpoint will be combined remission at week 12 defined as:

* 100% of the fistula tracts without any drainage by the external openings (occurring spontaneously or after gentle finger compression) And
* absence of collections >2 cm of the treated perianal fistulas confirmed by masked central MRI Patient requiring UST optimization will be considered in failure but will be followed until week 48

Secondary endpoints:

Definition

* Clinical remission: 100% of the fistula tracts without any drainage by the external openings (i.e, absence of any drainage by all fistula openings occurring spontaneously or after gentle finger compression)
* Clinical response (closure of at least 50% of all treated external openings that were draining at baseline)
* Radiological remission: absence of collections >2 cm of the treated perianal fistulas confirmed by masked central MRI
* Combined clinical and radiological remission at week 24 and 48.
* Clinical remission (i.e, absence of any drainage by all fistula openings occurring spontaneously or after gentle finger compression) at week 12, 24 and 48
* Absence of collections >2 cm of the treated perianal fistulas confirmed by masked central MRI at week 12, 24 and 48
* Evaluation of the magnetic resonance novel index for fistula imaging in CD at week 12, 24 and 48
* Clinical response (closure of at least 50% of all treated external openings that were draining at baseline) at week 12, 24 and 48
* Combined clinical response and radiological remission at week 48
* Perineal Disease Activity Index (PDAI), Crohn Disease Activity Index (CDAI) at week 12, 24 and 48
* Quality of life will be assessed with the Inflammatory Bowel Disease questionnaire (IBDQ) scores at week 24 and 48
* Correlation between response and remission and UST trough levels and antidrug (UST) antibodies at week 12, 24, 48
* Clinical response of UST optimization at week 48 (closure of at least 50% of all treated external openings that were draining at week 12)
* Clinical response at week 48 of UST introduction at W12 (closure of at least 50% of all treated external

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Adults with moderate to severe Crohn's disease for at least six months
* Patients with at least one active perianal fistula track (between the anus or low rectum and the perineum or vulva) confirmed by MRI within the previous 12 weeks
* Patients either naïve to anti-TNF therapy (50%) or refractory to anti-TNF therapy (50%).
* If female, subject is either not of child bearing potential, defined as post-menopausal for at least1 year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control during the study and for 150 days after the last dose:

  * Condoms, sponge and foam, jellies with diaphragm or intrauterine device (IUD). IUDs may fail during azathioprine treatment. Alternative or additional contraceptive measures are advised, if azathioprine is initiated
  * Oral or parenteral contraceptives for 3 months prior to study drug administration
  * A vasectomized partner
* Male subjects must agree to use an acceptable form of birth control, listed above at the start of azathioprine administration and for 90 days after last dose of azathioprine. Males should also commit to inform his partner(s) about it and to report any pregnancy to the investigator.
* If female, subject is not breast-feeding throughout the study and for 150 days after last dose.
* Subjects or his/her legal representative have voluntarily signed and dated an informed consent approved by and compliant with the requirements of this study protocol which has been approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)
* Adequate cardiac, renal and hepatic function as determined by the Principal Investigator and demonstrated by Screening laboratory evaluations, questionnaires and physical examination results that do not indicate an abnormal clinical condition which would place the subject at undue risk and thus preclude subject participation in the study
* Subject with a negative tuberculosis (TB) Screening Assessment [(including a Purified Protein Derivative (PPD) test < 5 mm and/or negative QuantiFERON-TB Gold test or equivalent and negative Chest X-Ray (CXR) (PA and lateral view)] at screening

Exclusion Criteria:

* Absence of written consent. People unable to give their consent (because of their physical or mental state)
* Pregnancy or breastfeeding
* Rectovaginal fistulas
* Rectal and/or anal stenosis
* Diverting stomas
* Abscess or collections >2 cm which are not properly drained ((i.e not drained at least 3 weeks before baseline and adequately treated provided that there is no anticipated need for any further surgery)
* History of colectomy.
* History of colonic mucosal dysplasia or adenomatous colonic polyps that are not removed.
* Screening stool trial positive for enteric pathogens or Clostridium difficile toxin. History of ongoing, chronic or recurrent infectious disease
* Positive HIV, Hepatitis B Virus (HBV),Hepatitis C Virus (HCV)
* Severe infection, chronic infection, history of recurrent infections, active infection including TB
* Malignancies or history of malignancies
* History of congestive heart failure (NYHA: Grade III and IV), demyelinating disease, current signs or history of severe/ progressive/uncontrolled renal, hepatic, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or systemic lupus erythematosus (SLE).
* History of transplanted organ, lymphoproliferative disease, any known malignancy
* Previous allergy immunotherapy for anaphylaxis, hypersensitivity to ustekinumab or to any excipients, or metronidazole or ciprofloxacin
* Previous use of a biologic agent targeting Interleukin 12 (IL12) and/or Interleukin 23 (IL 23), including but not limited to ustekinumab
* Oral corticosteroids at a dose > 40 mg prednisone or its equivalent per day at inclusion (oral steroids should be at stable dose at least 7 days before inclusion)
* Any current or previous use of the following within 8 weeks before the first trial agent injection : cyclosporine, tacrolimus, anti-TNF biologic agents or other agents intended to suppress or eliminate Tumor Necrosing Factor (TNF), and other biologics, including anti-integrin antibodies (approved or investigational), Janus Kinase (JAK) inhibitors (approved or investigational), or any current or previous use of an investigational agent
* Non-autologous stem cell therapy or biologic agents that deplete B or T cells <12 months prior to baseline
* Current or recent (less than 4 weeks) vaccination with attenuated live vaccines
* Patients using a prohibited medication
* Patients participating in another trial or being in a follow-up period for another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Combined clinical and radiological remission | Week 12
  Number of participants with 100% of the fistula tracts without any drainage by the external openings (occurring spontaneously or after gentle finger compression)
  - Number of participants with absence of collections >2 cm of the treated perianal fistulas confirmed by masked central MRI.

SECONDARY OUTCOMES:
Combined clinical and radiological remission | week 24 and week 48
  Number of participants with 100% of the fistula tracts without any drainage by the external openings (occurring spontaneously or after gentle finger compression)
  - Number of participants with absence of collections >2 cm of the treated perianal fistulas confirmed by masked central MRI.
Clinical response | week 12, week 24 and week 48
  Number of participants with closure of at least 50% of all treated external openings that were draining at baseline
MAGNIFI-CD26 | week 12, week 24 and week 48
  Evaluation of the magnetic resonance novel index for fistula imaging in CD (MAGNIFI-CD26)
PDAI | week 12, week 24 and week 48
  Perineal Disease Activity Index
IBDQ scores | week 24 and week 48
  Quality of life will be assessed with the Inflammatory Bowel Disease questionnaire scores
UST trough levels and antidrug | week 12 and week 24
  Correlation between response and remission and UST trough levels and antidrug (UST) antibodies
Clinical response of UST optimization | week 24 and week 48
  Number of participants with closure of at least 50% of all treated external openings that were draining at week 12
Clinical response of UST introduction at week 12 | week 24 and week 48
  Number of participants with closure of at least 50% of all treated external openings that were draining at week 12
CDAI | week 12, week 24 and week 48
  Crohn Disease Activity Index

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Rennes, Rennes, Brittany Region
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - CHU Clermont Ferrand, Clermont-Ferrand
  - APHP- Hopital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CHU Montpellier - St Eloi, Montpellier
  - Hôpital Hôtel Dieu, Nantes
  - CHU Nice- Hopital l'Archet, Nice
  - CHU Nîmes - Hôpital Universitaire Caremeau, Nîmes
  - Hôpital St Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Bichat, Paris
  - CHU LYON- Hopital Lyon Sud, Pierre-Bénite
  - CHU Roubaix, Roubaix
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - CHU de Tours - Hopital Trousseau, Tours
  - CHU Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993